CLINICAL TRIAL: NCT05942989
Title: The Effect of Reiki Applied to Pregnant Women in the Last Trimester on Breastfeeding Self-efficacy, Pregnancy Complaints and Quality of Life: A Randomized Controlled Study
Brief Title: The Effect of Reiki on Breastfeeding Self-efficacy, Pregnancy Complaints and Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Dilara Keklik, Research Assistant, PhD, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 134
Record Dates: First submitted 2023-06-23; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Obstetric Complication
Keywords: reiki; breastfeeding; self-efficiency; quality of life
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group that given education (Experimental): Reiki group
  Interventions: Other: Reiki implementation
- Control group (No Intervention): Group with no intervention

INTERVENTIONS:
Other: Reiki implementation — Reiki is implied by putting hands on the patient and it is believed that energy is transferred to patients by hands.
  Arms: Intervention group that given education

SUMMARY:
Despite the benefits of reiki application, no study has been found that examined the effects of reiki on breastfeeding self-efficacy, complaints during pregnancy and quality of life in pregnant women.

DETAILED DESCRIPTION:
Reiki, one of the complementary and alternative therapy (CAM) methods; It means "universal life energy" and is natural healing energy (Müller & Günther, 2006). This healing method is a way of treating others physically and spiritually (Vitale&O'Connor, 2006; Yücel, 2007). Reiki focuses on energy chakras and bio-psycho-spiritual healing. Reiki enables vital signs (blood pressure, pulse rate, respiratory rate) to reach normal levels, reduces acute and chronic pain, facilitates sleep, reduces anxiety and fear, relieves depression, reduces stress, provides relaxation, reduces the use of painkillers and increases coping skills. (Anderson & Ameling, 2001; Kelley & William, 2009; Lee et al., 2003; Pocotte & Salvador, 2008; Vitale, 2006).

Nurses are responsible for increasing the general health level of the mother by detecting and treating the existing diseases in the pregnant, providing timely diagnosis and treatment of potential problems that may arise, monitoring and evaluating the development of the mother and the fetus during pregnancy, giving care to the mother during pregnancy, general body care, nutrition, activity, family planning, It is responsible for providing information on signs of danger, care of the newborn and other issues that the mother may need, preparing the mother for birth physiologically and psychologically, thus increasing the quality of life of the mother (Taşkın, 2016).

ELIGIBILITY:
Inclusion Criteria:

First pregnancy In 28th and above gestational week Able to read and write Open to communication

Exclusion Criteria:

Having psychiatric history Diagnosed with risky pregnancy Having congenital anomaly in the baby in the postpartum period Having the childbirth preparation classes Receiving energy therapies before and having reiki training certificate

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 68 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Effect of reiki | starting from 28th gestational week until postpartum 6th week
  Reiki may affect breastfeeding self-efficacy and compliments in pregnancy

IPD SHARING:
Plan to Share IPD: No